CLINICAL TRIAL: NCT01374113
Title: An Open-label, Parallel-group, Single Center, Single Oral Dose Trial to Investigate the Pharmacokinetics (PK) of 50 mg Safinamide in Subjects With Moderate and Severe Renal Impairment Compared to Matched Subjects With Normal Renal Function
Brief Title: Safinamide Renal Impairment Trial
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Newron Pharmaceuticals SPA (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: EMR701165_025
Record Dates: First submitted 2011-06-14; First posted 2011-06-15 (Estimated); Last update posted 2013-03-29 (Estimated); Status verified 2011-10

CONDITIONS: Renal Impairment
Keywords: safinamide; pharmacokinetics; renal impairment; Moderate and Severe Renal Impairment
MeSH Terms: conditions — Renal Insufficiency; Lymphoma, Follicular | interventions — safinamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 1 (Experimental): Subjects with moderate renal impairment
  Interventions: Drug: 50mg safinamide
- Group 2 (Experimental): Subjects with severe renal impairment
  Interventions: Drug: 50mg safinamide
- Group 3 (Experimental): Matched subjects with normal renal function
  Interventions: Drug: 50mg safinamide

INTERVENTIONS:
Drug: 50mg safinamide — 50 mg safinamide on Day 1

SUMMARY:
The primary purpose of the trial is to investigate the pharmacokinetics (behaviour of the compound in the body) of safinamide in subjects with different degrees of renal impairment in comparison to matched subjects with normal renal function.

ELIGIBILITY:
Inclusion Criteria:

1. Renally impaired subjects - Subject with different degrees of renal impairment: moderate and severe renal impairment as assessed by Estimated Glomerular Filtration Rate (eGFR) according to Modification of Diet in Renal Disease (MDRD) equation at screening
2. Healthy subjects - Subject is in good age-appropriate physical and mental health as established by medical history, physical examination, electrocardiogram (ECG) and vital signs recordings, and results of biochemistry, haematology, coagulation and urinalysis testing within 3 weeks prior to dosing
3. All subjects have given written informed consent before any study-related activities are carried out

Exclusion Criteria:

1. Any other clinically relevant disease, condition, or therapy, which in the Investigator's opinion would exclude the subject from the trial, may pose a risk to the subject or interfere with the trial objectives.
2. Existence of surgical or medical condition, which, in the judgment of the Investigator, might interfere with the absorption, metabolism, or excretion of the drug and/or gastrointestinal motility
3. Renally impaired subjects - Acute renal failure of any etiology (including viral, toxic, or drug induced), renal transplantation within the previous 12 months, uncontrolled diabetes mellitus as judged by the Investigator, use of any drug affecting gastric acid secretion, such as proton pump inhibitors and antacids received within 48 hours prior to drug administration and for 24 hours after administration, Chronic heart failure (CHF) New York Heart Association (NYHA) class III and IV despite treatment at screening, change in used medication (prescribed by a physician or over-the-counter [OTC] medication) within 14 days prior to safinamide administration. Concomitant medication used for the treatment of renal impairment and accompanying diseases may be continued during the trial.
4. Healthy subjects - Use of any medication, including multi-vitamin preparations, received within 21 days prior to drug administration (or within six times the elimination half-life, whichever is longest), except combined oral contraceptives and occasional use of paracetamol or ibuprofen within 14 days before trial drug administration.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2011-06; Primary Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Cmax of safinamide in plasma in groups of subjects with different grades of renal function after a single dose of 50 mg safinamide | 12 to 14 days
AUC0-∞ of safinamide in plasma in groups of subjects with different grades of renal function after a single dose of 50 mg safinamide | 12 to 14 days

SECONDARY OUTCOMES:
Cmax of safinamide metabolite NW-1689 in plasma | 12 to 14 days
Cmax of safinamide metabolite NW-1153 in plasma | 12 to 14 days
Cmax of safinamide metabolite NW-1689 acylglucuronide in plasma | 12 to 14 days
AUC0-∞ of safinamide metabolite NW-1689 in plasma | 12 to 14 days
AUC0-∞ of safinamide metabolite NW-1153 in plasma | 12 to 14 days
AUC0-∞ of safinamide metabolite NW-1689 acylglucuronide in plasma | 12 to 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Anne Marquet, PharmaD, PhD, Study Director — Merck Serono S.A., Geneva
Locations (1):
- CRS Clinical Research Services Kiel GmbH, Kiel, Schleswig-Holstein, Germany